CLINICAL TRIAL: NCT00451633
Title: A Randomized, Double Blind, Placebo-Controlled Study To Investigate The Effect Of E2007 On Pharmacodynamic Responses To Levodopa Among Patients With Parkinson's Disease Who Experience Dyskinesia And Motor Fluctuations
Brief Title: The Effect Of E2007 On Pharmacodynamic Responses To Levodopa Among Patients With Parkinson's Disease Who Experience Dyskinesia And Motor Fluctuations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study group changed from patients to a healthy volunteers. A healthy-volunteer study is being planned to replace 213.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-E044-213
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

INTERVENTIONS:
Drug: E2007

SUMMARY:
A randomized, double blind, placebo-controlled study employing a mixed parallel group and fixed sequence cross-over design.

Patients will be randomized to one of two treatment groups ('E2007' or 'Placebo') in a 1:1 ratio and receive investigational drug treatment concomitant with their standard individualized anti-Parkinsonian therapy for a total of six weeks. Investigational drug treatment for patients in the E2007 treatment group will be started 2 mg E2007 o.d. but will be escalated to 4 mg E2007 o.d. after three weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will be eligible for the study if they meet all of the following inclusion criteria. Eligibility will be checked at screening and re-confirmed before the start of investigational drug dosing on Day -1 (ie, after completion and review of pre-dosing patient diaries and baseline assessments).

1. Men or women aged between 30 and 80 years, inclusive.
2. A diagnosis of idiopathic Parkinson's disease. Patients should fulfill the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria (Queen Square criteria) and have a rating of 2.4 on the Hoehn &Yahr scale when in an "off" state.
3. Receiving a regimen of anti-Parkinsonian treatments that has been optimized (according to the Investigator's opinion) and has been stable for at least four weeks before baseline. The regimen is not considered to be stable if 'as required' or 'on demand' dosing is routinely used or there is regular use of apomorphine or liquid forms of levodopa.
4. Taking levodopa at least three times during the waking day (not including bedtime or nighttime doses) and with a demonstrable response to each levodopa dose.
5. Consistently experiencing clinically-relevant, peak-effect levodopa-induced dyskinesias during the 'on' period following the morning dose of levodopa. Patients should:

   1. score .2 on Questions 32 and 33 of the full UPDRS at screening.
   2. have at least 3 h of 'on' time with dyskinesias on average per day recorded in the patient diary at baseline, of which 1 h is within the 4 h following the first morning dose of levodopa.
6. Consistently experiencing end-of-dose motor fluctuations. Patients should:

   1. score .1 on Question 39 of the full UPDRS at screening.
   2. have at least 1.5 h of 'off' time on average per day recorded in the patient diary at baseline.
7. Capable of adhering to the protocol requirements and providing written informed consent.

EXCLUSION CRITERIA:

Patients who meet any of the following exclusion criteria will not eligible for the study.

Eligibility will be checked at the Screening visit and re-confirmed before the start of investigational drug dosing on Day -1 (i.e., after completion and review of pre-dosing patient diaries and baseline assessments). All exclusion criteria must be observed.

1. A history of drug or alcohol abuse.
2. A history of suicide attempt or suicidal ideation within the past year.
3. Receiving antipsychotic treatment or a history of psychotic symptoms requiring antipsychotic treatment within the past year. Patients taking anti-depressant medications can enter the study providing the regimen is stable.
4. Receiving treatment with monoamine oxidase (MAO)-B inhibitors (e.g., selegiline, rasagiline).
5. Receiving treatment with medication known to induce CYP3A4 activity.
6. Receiving treatment with medications believed to have an effect on levodopa-induced dyskinesias (e.g., amantadine, dextromethorphan, clozapine, olanzapine, quetiapine).
7. Receiving treatment with medications known to exacerbate dyskinesias (eg, sodium valproate, CNS stimulants).
8. Failing to respond to the specified levodopa challenge, or where the levodopa challenge is not medically appropriate.
9. Experiencing dyskinesias unrelated to peak levodopa effect (e.g., "D-I-D" pattern).
10. Previous stereotactic surgery (e.g., pallidotomy, subthalamic nucleus deep brain stimulation) for Parkinson's disease.
11. Having received an investigational product within the four weeks leading up to Screening or having participated in a previous study with E2007.
12. Clinically significant cognitive impairment (mini-mental state examination [MMSE] <26 or fulfilling DSM IV criteria for dementia due to Parkinson's disease).
13. Active hepatic disease, significantly reduced hepatic function or significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper limit of the normal range).
14. Clinically significant ECG abnormalities, including prolonged QT interval (defined as QTc .450 msec).
15. Narrow-angle glaucoma.
16. Conditions affecting the peripheral or central sensory system that could interfere with pharmacodynamic evaluations of the effects of levodopa.
17. Women who are pregnant or lactating, or who are intending to become pregnant within two months of completion of the study.
18. Women of child-bearing potential who do not agree to use adequate non-hormonal contraception (e.g., intrauterine device, condoms with spermicide) throughout the study.
19. A history of drug hypersensitivity, especially hypersensitivity to any component of the investigational products or medication used for levodopa challenges.
20. A history of melanoma or suspicious, undiagnosed skin lesions.
21. Any condition that could, in the opinion of the Investigator, place the patient at increased risk or is likely to prevent completion of the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Levodopa pharmacokinetics will be assessed after each levodopa challenge. Blood samples for measurement of levodopa plasma
concentrations will be taken before and after levodopa dosing or until a full 'off' state is reached if earlier than 5 h.

SECONDARY OUTCOMES:
Pharmacodynamic assessments of dyskinesias and motor function; Goetz/Rush dyskinesia rating scale; modified abnormal involuntary movement scale (AIMS), and Unified Parkinson's disease rating scale motor examination sub-scale (UPDRS Part 3) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Nicotra, M.D., Ph.D., Study Director — Eisai Limited
Locations (5):
- Germany (3):
  - St. Josef Hospital, Bochum
  - Medizinische Hochschule Hannover, Hanover
  - Neurologische Universitatsklinik Marburg, Marburg
- Italy (2):
  - CESI - Centro Ricerche Cliniche - Fondazione Universita degli Studi, Chieti
  - U.O. Riabilitazione Neuromotoria, IRCCS San Raffaele Pisana, Roma